CLINICAL TRIAL: NCT03506243
Title: A Phase III, Multicenter, Blinded, Randomized, Controlled, Parallel, Comparative Study for the Evaluation of Safety and Efficacy of rhFSH Injection Compared With Gonal-F® Pen Undergoing Controlled Ovarian Hyper Stimulation IVF-ET
Brief Title: Randomized Controlled Study of Comparing Follitrope Versus Gonal-f in Chinese Infertility Women.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou YuYuan Bioscience Technology Co., Ltd. (Other)
Collaborators: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG1409CPL
Record Dates: First submitted 2018-04-11; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Infertility, Female
Keywords: IVF, rhFSH
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Test group (Experimental): Follitrope PFS
  Interventions: Biological: Follitrope PFS
- Control group (Active Comparator): Gonal-F pen
  Interventions: Biological: Gonal-f pen

INTERVENTIONS:
Biological: Follitrope PFS — Follitrope PFS
  Arms: Test group
Biological: Gonal-f pen — Gonal-f pen
  Arms: Control group

SUMMARY:
This study is for evaluating safety and efficacy of Recombinant human follicle-stimulating hormone (Follitrope) injection compared with Gonal-F® Pen undergoing controlled ovarian hyper stimulation in vitro fertilization - embryo transfer (IVF-ET) in China

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, blinded, randomized, controlled, parallel, comparative study for the evaluation of safety and efficacy of Recombinant human follicle-stimulating hormone injection (Follitrope) compared with Gonal-F® Pen undergoing controlled ovarian hyper stimulation in vitro fertilization - embryo transfer (IVF-ET) in China.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile adult women between 20 and 39 years at screening.
2. Infertile adult women with regular menstrual cycles of 25 to 35 days at screening.
3. Normal basal serum FSH, LH, E2, and P levels at the early follicular phase at screening.
4. If the cause of infertility is due to following reasons:

   * Tubal factor
   * Unknown reason
   * Male infertility
   * Combined factors
5. Willing to give voluntary written informed consent.

Exclusion Criteria:

1. Patients with a clinically significant systemic disease, endocrine or metabolic abnormalities.
2. Body Mass Index > 30 (BMI; kg/m2) at screening.
3. Patients with a uterine (fibroids (diameter greater than or equal to 2CM endometrium), endometrial polyps, intrauterine adhesions, uterine malformations), ovaries (polycystic ovary, ovarian cysts) or adnexa (hydrosalpinx) abnormalities at screening.
4. patients with uterine, ovarian surgery treatment
5. Patients who experienced of severe ovarian hyperstimulation symptoms (OHSS) in previous IVF cycles.
6. Patients who have shown poor response with gonadotropin hormone therapy.

   *At least two of the following three features must be present:

   ① A previous POR(≤3 retrieved oocyte with a conventional stimulation protocol)

   ② An abnormal ovarian reserve test (i.e. AFC < 5 follicles) at screening.
7. Abnormal metrorrhagia due to unknown reason at screening.
8. At least one of husband and wife to accept donor sperm or donor eggs or PGD subject
9. Subjects who are positive for HIV or syphilis at screening.
10. Significant known psychiatric disorder or who unable to understand the objectives and methods, etc. of this clinical trial and unable to comply with the study procedures at screening.
11. Presence of elicit alcohol, smoke or drug abuse habit at screening.
12. History of hypersensitivity to rhFSH or other pharmaceutical excipients of this drug.
13. Participation in any other clinical trial after registering for this study or have participated in another clinical study within 3 month before randomization in this study.
14. History of tumors of the ovary, breast, uterus, hypothalamus or pituary gland.
15. More than 3 times previously consecutive unsuccessful in vitro fertilization cycles at screening.
16. Subjects with no clomiphene citrate or gonadotropin treatment within 1 month before randomization.
17. Positive serum pregnancy test at screening.
18. 14 ± 2 days after the demotion, results of subjects who does not belong to the standard (antral follicle size ≥10mm)

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The total number of oocytes retrieved | 15 days after using FSH
  The total number of oocytes retrieved

SECONDARY OUTCOMES:
Total dose and duration of FSH administration | Throughout the study completion (e.g., 10 days)
  Total dose and duration of FSH administration
No. of follicles with diameter equal or more than 14 mm on hGH injection day | The day of hGH injection
  No. of follicles with diameter equal or more than 14 mm on hGH injection day
No. of embryo transferred | 3 days after the ovum pick-up
  No. of embryo transferred
Clinical pregnancy rate | 5 weeks after the embryo transfer
  Clinical pregnancy rate by g-sac
On-going pregnancy rate | 10 weeks after the embryo transfer
  On-going pregnancy rate by fetal heart-beat

CONTACTS AND LOCATIONS:
Overall Officials: Ying Pu Sun, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Hangzhou Yuyuan Bioscience Technology Co.,Ltd, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No